CLINICAL TRIAL: NCT00151905
Title: Nebulized Hypertonic Saline in the Treatment of Bronchiolitis in Infants
Brief Title: The Use of an Inhaled Salt Solution to Treat Viral Lung Infections in Infants.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sheikh Khalifa Medical City (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RC-09
Record Dates: First submitted 2005-09-07; First posted 2005-09-09 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2005-09

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; hypertonic saline
MeSH Terms: conditions — Bronchiolitis | interventions — Saline Solution, Hypertonic

INTERVENTIONS:
Drug: 3 % hypertonic saline

SUMMARY:
Bronchiolitis is a common viral lung infection in infants. Standard treatment often includes the use of inhaled medications which are usually first mixed with a standard salt solution. Inhalation of a more concentrated salt solution (hypertonic saline) has been successfully used to treat other types of lung disease in children and adults. The purpose of this study is to see if using inhaled hypertonic saline helps infants with bronchiolitis get better more quickly.

DETAILED DESCRIPTION:
Bronchiolitis is a common illness in infants and is associated with a significant morbidity. Standard therapy is controversial and largely ineffective; care is mostly supportive although nebulized medications continue to be commonly used. These medications are typically mixed with normal saline to produce a sufficient volume for efficient nebulization.

Inhaled hypertonic saline has been used to aid airway clearance in children with cystic fibrosis. It has also been used, in low dose, in two small studies in children with bronchiolitis. The current study is a randomized, double-blind, placebo-controlled, multi-center trial comparing frequent dosing with 3% hypertonic saline compared to normal saline in the treatment of infants hospitalized with bronchiolitis.

ELIGIBILITY:
Inclusion Criteria:

* Corrected age maximum 18 months, plus
* History of preceding viral upper respiratory tract infection, plus
* Presence of wheezing and/or crackles on auscultation, plus
* Respiratory Distress Assessment Instrument (RDAI) score of 4 or greater, or oxygen saturation of 93% or less in room air, plus
* Admitted to hospital

Exclusion Criteria:

* Prior history of wheezing, or
* History of chronic cardiopulmonary disease or immunodeficiency, or
* Critical illness at presentation requiring admission to ICU, or
* Use of nebulized hypertonic saline within previous 12 hours, or
* Prematurity (gestational age 34 weeks or less).

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-11; Study Completion 2006-09

PRIMARY OUTCOMES:
Length of stay.

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Kuzik, MD, FRCP, Principal Investigator — Sheikh Khalifa Medical City
Locations (3):
- Canada (2):
  - Victoria General Hospital, Victoria, British Columbia
  - Kingston General Hospital, Kingston, Ontario
- Sheikh Khalifa Medical City, Abu Dhabi, Abu Dhabi Emirate, United Arab Emirates